CLINICAL TRIAL: NCT03348488
Title: An Investigation of Transcapillary Plasma Refill During Ultrafiltration in Haemodialysis
Brief Title: Transcapillary Plasma Refill in Advanced Chronic Kidney Disease
Acronym: PRUf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); Manchester Metropolitan University (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R04305
Record Dates: First submitted 2017-08-21; First posted 2017-11-21 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Haemodynamic Instability

STUDY DESIGN:
Intervention Model Description: The 2 arms applied to the same subject studied twice (case controlled)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard ultrafiltration (No Intervention): standard ultrafiltration (fluid removal from the body by dialysis at the prescribed volume and rate) during a conventional treatment
- High dose ultrafiltration (Active Comparator): Intervention= Fixed rate high dose ultrafiltration (fluid removed from the body by dialysis) of 1 litre per hour over 1 hr instaed of standard ultrafiltration rate and volume.
  Interventions: Procedure: Ultrafiltration dose

INTERVENTIONS:
Procedure: Ultrafiltration dose — Fixed high volume of ultrafiltration over an hour during dialysis
  Other Names: Ultrafiltration rate
  Arms: High dose ultrafiltration

SUMMARY:
Background: Haemodynamic instability during haemodialysis has long been linked to poor cardiovascular outcomes. It does not always reflect overall hydration but rather plasma volume depletion, with a delay in plasma refill from other body compartments, and vasodilatation, mediated by endothelial factors. Our understanding of these processes remains largely incomplete. Despite our ability to monitor relative blood volume during haemodialysis our knowledge concerning the factors affecting plasma refill remain incomplete. This may be due to variations observed between individuals. Understanding the pattern of fluid shifts variation between the different body compartment and the factors affecting these behaviours in different individuals or at different hydration states could be a vital component of our management of intradialytic haemodynamic instability but also overhydration.

Aims and Objectives: The aim of this study is to describe plasma refill rate, during haemodialysis using a non-invasive, continuous, real-time data capture during ultrafiltration. The study will attempt to describe different refilling phenotypes in the study population and seek association with biochemical and haematological parameters linked to variability in refilling rates.

Methodology: This study will attempt to describe variations in the plasma refill rate of prevalent dialysis patients during their normal haemodialysis treatment and during a session of 3 hours of haemodialysis preceded by 1 hour of isolated ultrafiltration using the in-built blood volume monitoring module of their haemodialysis machine and the TMON software that collects continuous, real-time data by interfacing with the computer network. To achieve this, a bolus of 100-300ml of intravenous dialysis replacement fluid will be administered at the beginning of each of the 2 studied sessions.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent haemodialysis patient at CMFT and satellite units

Exclusion Criteria:

* Withdrawal of consent.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Plasma refilling rate | Continuous derivation of the refilling rate during a four hour haemodialysis treatment
  To assess absolute plasma volume changes during ultrafiltration on haemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Mitra, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No